CLINICAL TRIAL: NCT03836898
Title: Presbyopic Phakic Intraocular Lens for Myopia Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gemini Eye Clinic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PhakicIOL Presbyopia
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Presbyopia; Myopia
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation phakic intraocular lens (Experimental): Presbyopic posterior chamber phakic intraocular lens IPCL implanted to the participants eye
  Interventions: Device: Presbyopic posterior chamber phakic intraocular lens IPCL

INTERVENTIONS:
Device: Presbyopic posterior chamber phakic intraocular lens IPCL — Presbyopic posterior chamber phakic intraocular lens IPCL (EyeolUK, United Kingdom) has a refractive optic and diffractive trifocal pattern on its anterior optical surface to correct both distance and near refractive errors. Presbyopic addition is manufactured in a range of +1.0 to + 4.0 diopters (D) in 0.5 D steps.

SUMMARY:
This is a prospective single-center study of implantations of the presbyopic version of phakic intraocular lens IPCL (EyeolUK, United Kingdom).

DETAILED DESCRIPTION:
Participants are impanted with the phakic intraocular lens IPCL (EyeolUK, United Kingdom) and monitored during 2 years period. Visual acuity for near and distance is evaluated, along with refraction and endothelium cell density.

ELIGIBILITY:
Inclusion Criteria:

* CDVA < 0.3 LogMAR
* Presbyopia with moderate to high myopia
* Phakic

Exclusion Criteria:

* Corneal endotehleial cell density below 2000 cells/mm2
* Corneal dystrophies
* ACD less than 2.8 mm
* history or current uveitis
* acute ocular inflammation
* glaucoma
* chronic uveitis
* previous intraocular or refractive surgery
* preexisting ocular pathologic which may affect postoperative results

Ages: 38 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Uncorrected Distance Visual Acuity (UDVA) | 2 years
  Distance visual acuity tested without any correction
Change in Uncorrected Near Visual Acuity (UNVA) | 2 years
  Near visual acuity tested without any correction

SECONDARY OUTCOMES:
Change in Corrected Distance Visual Acuity (CDVA) | 2 years
  Distance visual acuity tested with correction
Change in Corrected Near Visual Acuity (CNVA) | 2 years
  Near visual acuity tested with correction
Change in distance refraction | 2 years
  Expressed as spherical equivalent sp.Eq (D)
Change in near refraction | 2 years
  Expressed as spherical equivalent sp.Eq (D)

CONTACTS AND LOCATIONS:
Locations (1):
- Gemini Eye Clinic, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stodulka P, Slovak M, Sramka M, Polisensky J, Liska K. Posterior chamber phakic intraocular lens for the correction of presbyopia in highly myopic patients. J Cataract Refract Surg. 2020 Jan;46(1):40-44. doi: 10.1097/j.jcrs.0000000000000033. PMID 32050231